CLINICAL TRIAL: NCT03624478
Title: A Pilot/Phase II Trial of Hypofractionated Radiotherapy to the Whole Breast Alone Before Breast Conserving Surgery
Brief Title: Hypofractionated Radiation Therapy in Treating Participants With Breast Cancer Before Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1732; NCI-2018-01606 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1732 (Other: Mayo Clinic in Arizona); 17-004130 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2018-08-06; First posted 2018-08-10 (Actual); Results first posted 2022-12-15 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8
MeSH Terms: interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (hypofractionated radiation therapy) (Experimental): Participants undergo hypofractionated radiation therapy daily for 5 days, then undergo standard of care surgery 4-16 weeks after radiation therapy.
  Interventions: Radiation: Hypofractionated Radiation Therapy

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated Radiotherapy; hypofractionation

SUMMARY:
This phase II trial studies how well hypofractionated radiation therapy works in treating participants with breast cancer before surgery. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the pathologic complete response (pCR) rate after hypofractionated radiotherapy to the whole breast alone, based on the postsurgical specimen.

SECONDARY OBJECTIVES:

I. To evaluate acute and late toxicity with preoperative radiation including grade >= 2 pneumonitis.

II. To estimate the 5-year locoregional control, distant recurrence, invasive disease-free survival, cause-specific survival, and overall survival.

CORRELATIVE AND EXPLORATORY OBJECTIVES:

I. To evaluate patient-reported outcomes. II. To evaluate clinical features, treatment technique, dose-volume parameters, histologic and genetic variants associated with adverse events, and fair and poor cosmetic outcomes or unplanned surgical intervention.

III. Evaluate tumor mutation signatures before and after radiation; correlate tumor mutation signatures before and after radiation with pathologic information at the time of surgery.

IV. To describe the pathologic changes seen in breast cancer patients with preoperative radiation.

OUTLINE:

Participants undergo hypofractionated radiation therapy daily for 5 days, then undergo standard of care surgery 4-16 weeks after radiation therapy.

After completion of study treatment, participants are followed up at 12 weeks, 6, 12, 24, and 36 months, and 5 years after radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of breast cancer
* Clinical stage T0-T2 N0 M0
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 to 2
* Able to and provides Institutional Review Board (IRB) approved study specific written informed consent
* Study entry must be within 120 days of last biopsy (breast)
* Able to complete all mandatory tests
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Planned breast surgery and indications for whole breast radiotherapy

Exclusion Criteria:

* Medical contraindication to receipt of radiotherapy
* Severe active co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or providing informed consent
* Active systemic lupus or scleroderma
* Pregnancy
* Women of childbearing potential who are unwilling to employ adequate contraception
* Prior receipt of ipsilateral breast or chest wall radiation
* Recurrent breast cancer
* Indications for comprehensive regional nodal irradiation
* No neo-adjuvant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2025-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E. Vargas, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (hypofractionated radiation therapy): Participants undergo hypofractionated radiation therapy daily for 5 days, then undergo standard of care surgery 4-16 weeks after radiation therapy.>>
  >> Hypofractionated Radiation Therapy: Undergo hypofractionated radiation therapy
Period: Overall Study
Arm/Group | Treatment (hypofractionated radiation therapy)
Started | 25
Completed | 24
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Hypofractionated Radiation Therapy)
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Enrollment Site [Count of Participants; unit: Participants]
  Arizona | 16
  Florida | 8
Method of Payment [Count of Participants; unit: Participants]
  Medicare | 9
  Private Insurance | 15

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR) Rate Defined as a Residual Tumor Burden of 0-1 in the Surgical Specimen
Description: The proportion of successes (number of patients achieving pCR at time of definitive surgery) will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.
Time Frame: up to 2 years
Population: If more than the target number of 22 patients are accrued, the additional patients will not be used to evaluate the stopping rule or used in any decision making process.
Measure: Number; unit: proportion of participants
Groups:
- Treatment (hypofractionated radiation therapy): Participants undergo hypofractionated radiation therapy daily for 5 days, then undergo standard of care surgery 4-16 weeks after radiation therapy.
  >>
  >> Hypofractionated Radiation Therapy: Undergo hypofractionated radiation therapy
Arm/Group | Treatment (hypofractionated radiation therapy)
Number analyzed (Participants) | 22
proportion of participants | 0.64

2. Secondary Outcome: Number of Participants With Acute Adverse Events (AE)
Description: The maximum grade for each type of acute AE will be recorded for each patient. Data will be summarized as frequencies and relative frequencies. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.
Time Frame: Up to 180 days post radiation therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (hypofractionated radiation therapy)
Number analyzed (Participants) | 24
Participants
  Any Grade 2+ AE: No | 16
  Any Grade 2+ AE: Yes | 8
  Any Grade 3+ AE: No | 19
  Any Grade 3+ AE: Yes | 5

3. Secondary Outcome: Incidence of Late Adverse Events
Description: The maximum grade for each type of late AE will be recorded for each patient. Data will be summarized as frequencies and relative frequencies by treatment arm. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.
Time Frame: Up to 5 years post radiation therapy
Reporting Status: Not Posted

4. Secondary Outcome: Locoregional Control
Description: The cumulative incidence of locoregional recurrence will be estimated using a competing risks method (Gooley et al.). The competing risks will be distant breast cancer recurrence and death.
Time Frame: Up to 5 years
Reporting Status: Not Posted

5. Secondary Outcome: Invasive Disease-free Survival
Description: Will be estimated with a Kaplan-Meier estimator and curve. Estimates will be given for specific time points along with 95% confidence intervals (CIs).
Time Frame: From registration until the time of disease recurrence or death due to any cause, assessed up to 5 years
Reporting Status: Not Posted

6. Secondary Outcome: Distant Recurrence
Time Frame: Up to 5 years
Reporting Status: Not Posted

7. Secondary Outcome: Disease- Free Survival
Description: Will be estimated with a Kaplan-Meier estimator and curve. Estimates will be given for specific time points along with 95% CIs.
Time Frame: From registration until the time of disease recurrence or death due to any cause, assessed up to 5 years
Reporting Status: Not Posted

8. Secondary Outcome: Cause-specific Survival
Description: as for outcome 7
Time Frame: From registration to death due to breast cancer assessed up to 5 years
Reporting Status: Not Posted

9. Secondary Outcome: Overall Survival
Description: as for outcome 7
Time Frame: From registration to death due to any cause assessed up to 5 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Patient Self-reporting of Toxicities
Description: The subscales of the Breast Cancer Treatment Outcomes Scale (BCTOS), elements from Patient Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE), and other patient reported measures such as fatigue, breast pain, breast shape, and arm related morbidity outlined in the appendix will be summarized as the mean +/- SD and median (minimum value, maximum value). Scale score trajectories over time will be examined using stream plots and mean plots with standard deviation error bars overall. Analysis will include percent change from baseline using t-tests and generalized linear models to test for changes at each time point and non-zero slope respectfully.
Time Frame: Up to 5 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Patient Self-reported Cosmetic Outcomes
Description: Assessed using a modified Harvard Cosmesis Scale and the BCTOS. The values of the cosmesis instruments (patient self-reported and panel-assessed) will be summarized with the frequencies and confidence intervals of fair or poor cosmesis events.
Time Frame: Baseline up to 5 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Panel Assessed Cosmetic Outcome
Description: Cosmesis will be assessed by a panel of breast cancer medical providers using digital photographs.
Time Frame: Baseline up to 2 years
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Clinical Features, Treatment Technique, Dose-volume Parameters, Histologic and Genetic Variants
Description: Associated with adverse events, and fair and poor cosmetic outcomes or unplanned surgical intervention.
Time Frame: Up to 5 years
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Tumor Mutation Signatures
Description: Will be analyzed before and after radiotherapy as compared to pathologic information at the time of surgery. Continuous variable will be compared using unpaired t tests and nominal variables will be compared using contingency tables and Chi square analyses.
Time Frame: Up to 5 years
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Pathologic Changes Seen in Breast Cancer Patients With Preoperative Radiation
Description: Will be described.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 3 years
Arm/Group | Treatment (hypofractionated radiation therapy)
All-Cause Mortality (participants affected / at risk) | 2/24
Serious Adverse Events (participants affected / at risk) | 2/24
Other Adverse Events (participants affected / at risk) | 22/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (hypofractionated radiation therapy) (N=24)
Death NOS (General disorders and administration site conditions) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (hypofractionated radiation therapy) (N=24)
Pain (General disorders and administration site conditions) | 17 (39)
Dermatitis radiation (Injury, poisoning and procedural complications) | 12 (16)
Seroma (Injury, poisoning and procedural complications) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 4 (9)
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 7 (17)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 11 (22)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Lymphedema (Vascular disorders) | 8 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT03624478/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT03624478/ICF_001.pdf